CLINICAL TRIAL: NCT06625567
Title: Effect of Preoperative Patient Education Via Animated Videos on Anxiety in Patients Undergoing Hysteroscopy Without Anesthesia
Brief Title: The Effect of Preoperative Animated Videos on Anxiety in Patients Undergoing Hysteroscopy Without Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Neta Eisenberg Kogan, Attending physician in the gynecology endoscopy unit, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11-23
Record Dates: First submitted 2024-09-27; First posted 2024-10-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A prospective, non-blinded, randomized comparative study including patients undergoing hysteroscopy without anesthesia in the outpatient hysteroscopy clinic at Shamir (Assaf Harofe) medical center. In the control group, patients will receive the standard education regarding the procedure. In the study group, patients will also watch a short educational video.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients undergoing hysteroscopy without anesthesia. Patients will receive the standard education regarding the procedure.
- Intervention group (Experimental): Patients undergoing hysteroscopy without anesthesia. Patients will receive the standard education regarding the procedure and will also watch a short educational video.
  Interventions: Other: Animated video

INTERVENTIONS:
Other: Animated video — Patients will watch an educational video describing the procedure before hysteroscopy without anesthesia
  Arms: Intervention group

SUMMARY:
Office hysteroscopy is a gynecologic procedure performed to evaluate the uterine cavity. In the majority of cases, this procedure is performed without anesthesia.

Previous studies found significant levels of anxiety in women undergoing this procedure. In the current study, we will assess if the use of a preoperative audiovisual animated video describing will affect patient's anxiety and pain.

All patients will receive the standard education regarding the procedure from the physician. In the study group, in addition, an educational animated video will be shown. Subsequently, all patients will be asked to fill an anxiety assessment questionnaire in Hebrew (State-Trait Anxiety Inventory - State). After the procedure, patients will be asked about their pain level (VAS). Finally, patients in the study group will be asked to fill a short questionnaire regarding the educational video.

DETAILED DESCRIPTION:
Backgroung: Office hysteroscopy is a gynecologic procedure performed to evaluate the uterine cavity in cases of various gynecologic problems and abnormal ultrasound findings (such as endometrial polyps, fibroids, abnormal uterine bleeding, and infertility). In the majority of cases, this procedure is performed without anesthesia using a small diameter (~3-4 mm) fibro-optic equipment and a minimally invasive "no-touch" vaginoscopic technique. Although this procedure is considered to be non-painful and well tolerated, previous studies found significant levels of anxiety in women undergoing hysteroscopy without anesthesia. Several non-pharmacologic approaches have been suggested with the aim of decreasing patients' anxiety. Among those, communication and patient's education appear to have a significant role. In the current study, we will assess the effect of an educational video describing the procedure on patients' anxiety before hysteroscopy without anesthesia, and compare it to the anxiety levels of patients who received the standard education.

Objective To assess if the use of a preoperative audiovisual animated video describing hysteroscopy without anesthesia will affect patient's anxiety and pain.

Design A prospective, non-blinded, randomized comparative study including patients undergoing hysteroscopy without anesthesia in the outpatient hysteroscopy clinic at Shamir (Assaf Harofe) medical center. In the control group, patients will receive the standard education regarding the procedure. In the study group, patients will also watch a short educational video.

Inclusion criteria:

Adult patients (≥18 years) undergoing hysteroscopy without anesthesia in the hysteroscopy outpatient clinic.

Exclusion criteria:

1. Patients who are unable to understand or watch the audiovisual video
2. Patients who are unable to understand or to complete the Hebrew questionnaires. The study will include a total of 200 patients. The patients will be randomly assigned to the study or to the control group according to the day of the procedure (i.e., on select pre-determined days all patients will be assigned either to the control group or to the study group).

All patients will receive the standard education regarding the procedure from the physician. In the study group, in addition, an educational animated video will be shown. Subsequently, all patients will be asked to fill an anxiety assessment questionnaire in Hebrew (State-Trait Anxiety Inventory - State) (Appendix 1). The hysteroscopy will be performed according to the routine clinical care. After the procedure, patients will be asked about their pain level (VAS). Finally, patients in the study group will be asked to fill a short questionnaire regarding the educational video (Appendix 2).

Demographic variable (age, body mass index, obstetrical history and gynecologic history) will be also collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) undergoing hysteroscopy without anesthesia in the hysteroscopy outpatient clinic.

Exclusion Criteria:

* Patients who are unable to understand or watch the audiovisual video
* Patients who are unable to understand or to complete the Hebrew questionnaires.
* Age < 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2023-02-26 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Anxiety levels before the procedure | Immediately before procedure
  Anxiety levels before the procedure will be assesses according to the State-Trait Anxiety Inventory - State questionnaire which is composed out of 20 questions. Scoring is 1-4 for each question and total score is calculated using a formula with a final score of under 30 indicating low anxiety, 31-45 moderate anxiety and 46 and above high level of anxeity . The hysteroscopy will be performed according to the routine clinical care.

SECONDARY OUTCOMES:
Pain levels after procedure | Immediately after procedure
  Pain levels measure by Visual Analogue Scale scored from 0-10 (0 indicating no pain and 10 the highest level of pain) after procedure is done

CONTACTS AND LOCATIONS:
Overall Officials: Neta Eisenberg Kogan, Principal Investigator — Shamir Assaf Harofeh medical center
Locations (1):
- Shamir medical center, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: Yes
The data that is collected will be shared
Supporting Information: CSR
Time Frame: The data will be shared onced sent to publication for unlimited time
Access Criteria: The data will be published in suitable journals for that purpose

REFERENCES:
- [Result] Angioli R, De Cicco Nardone C, Plotti F, Cafa EV, Dugo N, Damiani P, Ricciardi R, Linciano F, Terranova C. Use of music to reduce anxiety during office hysteroscopy: prospective randomized trial. J Minim Invasive Gynecol. 2014 May-Jun;21(3):454-9. doi: 10.1016/j.jmig.2013.07.020. Epub 2013 Aug 17. PMID 23962572
- [Result] Carta G, Palermo P, Marinangeli F, Piroli A, Necozione S, De Lellis V, Patacchiola F. Waiting time and pain during office hysteroscopy. J Minim Invasive Gynecol. 2012 May-Jun;19(3):360-4. doi: 10.1016/j.jmig.2012.01.017. Epub 2012 Mar 3. PMID 22387163
- [Result] Vitale SG, Caruso S, Ciebiera M, Torok P, Tesarik J, Vilos GA, Cholkeri-Singh A, Gulino FA, Kamath MS, Cianci A. Management of anxiety and pain perception in women undergoing office hysteroscopy: a systematic review. Arch Gynecol Obstet. 2020 Apr;301(4):885-894. doi: 10.1007/s00404-020-05460-2. Epub 2020 Mar 5. PMID 32140807
- [Result] Gambadauro P, Navaratnarajah R, Carli V. Anxiety at outpatient hysteroscopy. Gynecol Surg. 2015;12(3):189-196. doi: 10.1007/s10397-015-0895-3. Epub 2015 May 13. PMID 26283891